CLINICAL TRIAL: NCT06017999
Title: A Randomized, Double-Blind, Placebo Controlled Trial to Evaluate the Safety and Efficacy of XG005 Tablets in Subjects Undergoing Bunionectomy
Brief Title: XG005 for Pain Control in Subjects Undergoing Bunionectomy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Xgene Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PR-XG005-02-BUN-01
Record Dates: First submitted 2023-08-18; First posted 2023-08-30 (Actual); Results first posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- high dose (Experimental): XG005 1250 mg Q12 hours
  Interventions: Drug: XG005 tablet
- low dose (Experimental): XG005 750 mg Q12 hours
  Interventions: Drug: XG005 tablet; Drug: Placebo tablet
- placebo (Placebo Comparator): placebo Q12 hours
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: XG005 tablet — Subjects will receive XG005 prior to surgery and every 12 hours for 72 hours.
  Arms: high dose; low dose
Drug: Placebo tablet — Subjects will receive placebo prior to surgery and every 12 hours for 72 hours.
  Arms: low dose; placebo

SUMMARY:
This study will evaluate the safety, efficacy, and PK of low dose (750 mg) and high-dose (1250 mg) XG005 oral tablets compared with placebo in subjects undergoing bunionectomy. Subjects will be confined in the clinic from check-in through 72 hours post-surgery to monitor subject safety.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, parallel-group, placebo-controlled study. Eligible subjects will be randomized in a 1:1:1 ratio to receive either 750 mg XG005, 1250 mg XG005, or placebo, twice a day, post bunionectomy surgery in domiciled clinic. Subjects and all study staff performing study assessments will be blinded to treatment allocation. Subjects will be discharged at a reasonable hour of the day after the end of the 72-hour treatment period.There will be a Follow-up Visit on Day 15.

ELIGIBILITY:
Main inclusion criteria:

* Scheduled to undergo unilateral first metatarsal bunionectomy
* Have negative urine drug screen
* Non-pregnant, non-lactating

Main exclusion criteria:

* Medical condition or history that in the investigator's opinion could adversely impact the subject's participation or safety
* Use of disallowed medications (e.g. pain medication, CNS active drugs such as benzodiazepines, tricyclic antidepressants, Serotonin, and norepinephrine reuptake inhibitors (SNRIs), selective serotonin reuptake inhibitors (SSRIs), or any other serotonergic medications, parenteral or oral corticosteroids)
* Antihypertensive agent or diabetic regimen at a dose that has not been stable for at least 30 days
* Digoxin, warfarin lithium, theophylline preparations, aminoglycosides, and all antiarrhythmics
* Monoamine oxidase inhibitors (MAOIs)
* Positive HbsAg and/or anti-HBc but negative anti-HBs
* HIV infection
* History of illicit drug use
* History of opioid dependence
* History of NSAID-induced bronchospasm or presence of nasal polyps, history of asthma or chronic rhinitis
* Significant history of allergic reactions or known intolerance to naproxen, pregabalin or any gabapentinoid, or to any rescue medication used in the study, or any medication used in the surgical and anesthetic protocol.
* Presence of severe depression as indicated by Patient Health Questionnaire (PHQ 9) total score of ≥20 or item 9 score >0
* Presence of severe anxiety as indicated by General Anxiety Disorder (GAD-7) score of ≥15
* Presence of history of suicidal behavior or ideation as indicated by the C-SSRS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Arizona Research Center, Phoenix, Arizona
  - Pacific Research Network, San Diego, California
  - Clinical Pharmacology of Miami, Hialeah, Florida
  - Midwest Clinical Research Center, Dayton, Ohio
  - First Surgical Hospital, Bellaire, Texas
  - Legent Orthopedic Hospital, Carrollton, Texas
  - Memorial Hermann Village, Houston, Texas
  - Endeavor Clinical Trials, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High dose | Low dose | Placebo
Started | 152 | 149 | 149
Safety set (The Safety Population was defined as all subjects who received study medication. Subjects were analyzed according to the actual treatment they received.) | 152 | 149 | 147
Completed | 148 | 142 | 135
Not Completed | 4 | 7 | 14
Not completed — Withdrawal by Subject | 0 | 4 | 3
Not completed — Adverse Event | 2 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Non-Compliance | 0 | 0 | 1
Not completed — Lack of Efficacy | 1 | 0 | 7
Not completed — COVID Positive | 0 | 1 | 0
Not completed — Did Not Disclose Amount of EtOH Consumed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population was defined as all randomized subjects (Intend-To-Treat population).
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose | Low Dose | Placebo | Total
Number analyzed (Participants) | 152 | 149 | 149 | 450
Age, Categorical [Count of Participants; unit: Participants] — The number of participants met the protocol requirement regarding the participants to be male or female, aged 18-80 years.
  Participants
    <=18 years | 1 | 1 | 1 | 3
    Between 18 and 65 years | 146 | 140 | 137 | 423
    >=65 years | 5 | 8 | 11 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 117 | 120 | 360
  Male | 29 | 32 | 29 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — The number of participants from various ethnic backgrounds.
  Participants
    Hispanic or Latino | 57 | 50 | 57 | 164
    Not Hispanic or Latino | 95 | 97 | 91 | 283
    Unknown or Not Reported | 0 | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — The number of participants from various races.
  Participants
    American Indian or Alaska Native | 0 | 1 | 0 | 1
    Asian | 5 | 2 | 1 | 8
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
    Black or African American | 40 | 55 | 49 | 144
    White | 103 | 82 | 94 | 279
    More than one race | 2 | 1 | 0 | 3
    Unknown or Not Reported | 2 | 7 | 5 | 14
Region of Enrollment [Count of Participants; unit: Participants] — The number of participants from the US.
  Participants
    United States | 152 | 149 | 149 | 450
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI) was assessed as part of eligibility screening. Participants were required to have a body weight greater than 50 kg and a BMI less than 39 kg/m² to meet the inclusion criteria. BMI was calculated as weight in kilograms divided by height in meters squared (kg/m²). Population: Three participants in the Placebo group had their BMI data not captured.
  kg/m^2
    number analyzed (Participants) | 152 | 149 | 146 | 447
    (all) | 28.37 (4.370) | 28.52 (4.464) | 28.05 (4.764) | 28.32 (4.527)

OUTCOME MEASURES:

1. Primary Outcome: Compared the Summed Pain Intensity From the End of Surgery to 48 Hours (SPI48) Between the High-dose XG005 Group and the Placebo Group Postoperatively.
Description: The primary efficacy endpoint compared the Summed Pain Intensity from the End of Surgery to 48 Hours (SPI48) between the high-dose XG005 group and the placebo group postoperatively.
  Subject-reported pain assessments via a standard 11-point Numeric Pain Rating Scale (NPRS, a scale of 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, and 10). 0 means "no pain",10 means "worst pain imaginable") at the following time points post-end of surgery: 0, 1, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24, 30, 36, 42, 48 hours within a ±10-minute window.
  Each pairwise treatment comparison (e.g., high dose vs. placebo, low dose vs. placebo) was analyzed using a separate ANCOVA model that included only the relevant treatment arms and adjusted for study site. As a result, the placebo least squares mean may differ slightly across comparisons due to differences in covariate adjustment.
  For the high-dose versus placebo comparison, SPI48 ranged from 0 to 425 in the high-dose group and from 0 to 446 in the placebo group.
Time Frame: SPI NPRS collection times occurred at 0, 1, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24, 30, 36, 42, 48 hours, within a ±10-minute window.
Measure: Least Squares Mean (Standard Error); unit: Numeric score
Arm/Group | High dose | Placebo
Number analyzed (Participants) | 152 | 149
Numeric score | 132.63 (8.004) | 285.99 (8.183)
Statistical Analysis 1: Comparison: High dose vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least Square Mean (LSM) difference = -153.35, 95% CI 2-sided [-173.80 to -132.91]

2. Secondary Outcome: Compared the Summed Pain Intensity From the End of Surgery to 48 Hours (SPI48) Between the Low-dose XG005 Group and the Placebo Group Postoperatively.
Description: The secondary efficacy endpoint compared the Summed Pain Intensity from the End of Surgery to 48 Hours (SPI48) between the low-dose XG005 group and the placebo group postoperatively.
  Subject-reported pain assessments via a standard 11-point Numeric Pain Rating Scale (NPRS, a scale of 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, and 10). 0 means "no pain",10 means "worst pain imaginable") at the following time points post-end of surgery: 0, 1, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24, 30, 36, 42, 48 hours within a ±10-minute window.
  The pairwise treatment comparison was analyzed using a separate ANCOVA model that included only the relevant treatment arms and adjusted for study site. As a result, the placebo least squares mean may differ slightly across comparisons due to differences in covariate adjustment.
  For the low-dose versus placebo comparison, SPI48 ranged from 0 to 383 in the low-dose group and from 0 to 446 in the placebo group.
Time Frame: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Numeric score
Arm/Group | Low dose | Placebo
Number analyzed (Participants) | 149 | 149
Numeric score | 157.86 (8.345) | 289.50 (8.500)
Statistical Analysis 1: Comparison: Low dose vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least Square Mean (LSM) difference = -131.64, 95% CI 2-sided [-153.13 to -110.16]

ADVERSE EVENTS:
Time Frame: The AE reporting period began at the time of the first dose of the study drug and ended 30 days after the last dose of the study drug, up to five weeks. AEs starting after the administration of the first dose of the study medications were considered to be TEAEs. All AEs were followed until they were resolved, stable, or deemed by the investigator to be not clinically significant, over a maximum period of five weeks.
Arm/Group | High dose | Low dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/152 | 0/149 | 0/147
Serious Adverse Events (participants affected / at risk) | 0/152 | 0/149 | 0/147
Other Adverse Events (participants affected / at risk) | 88/152 | 69/149 | 62/147
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High dose (N=152) | Low dose (N=149) | Placebo (N=147)
Somnolence (Nervous system disorders) | 23 (25) | 16 (16) | 0 (0)
Dizziness (Nervous system disorders) | 21 (22) | 17 (19) | 6 (7)
Nausea (Gastrointestinal disorders) | 24 (27) | 16 (18) | 19 (19)
Constipation (Gastrointestinal disorders) | 18 (18) | 13 (13) | 7 (7)
Vomitting (Gastrointestinal disorders) | 9 (11) | 5 (6) | 6 (6)
Headache (Nervous system disorders) | 7 (7) | 8 (9) | 12 (15)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 3 (4) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 5 (5)
Vision blurred (Eye disorders) | 5 (5) | 3 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Diplopia (Eye disorders) | 4 (4) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Upon study completion, the sponsor decides data reporting, publication venue, and authorship. Data remain the sponsor's property and require sponsor approval for publication, which will not be unreasonably withheld.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/99/NCT06017999/Prot_SAP_000.pdf